CLINICAL TRIAL: NCT02234089
Title: Therapy Pathways in the Treatment of Hormone Naïve Prostate Cancer Patients With and Without Comorbidities Treated With Degarelix or Luteinizing-Hormone-Releasing-Hormone (LHRH) Agonists.
Acronym: ProComD
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000156
Record Dates: First submitted 2014-08-20; First posted 2014-09-09 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Advanced Prostate Cancer
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Degarelix
  Interventions: Drug: Degarelix
- LHRH agonist
  Interventions: Drug: LHRH agonist (Leuprorelinacetat, Goserelinacetat, Buserelinacetat, Triptorelinacetat)

INTERVENTIONS:
Drug: Degarelix — According to medical practice
  Other Names: Firmagon®
  Groups: Degarelix
Drug: LHRH agonist (Leuprorelinacetat, Goserelinacetat, Buserelinacetat, Triptorelinacetat) — According to medical practice
  Groups: LHRH agonist

SUMMARY:
The purpose of this study is to detect factors influencing decision making for treatment pathways of hormone-naïve prostate cancer patients with and without comorbidities receiving medicinal androgen deprivation therapy (Degarelix or LHRH agonists).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Prostate Cancer and indicated for ADT according to Summary of Product Characteristics (SmPC)
* Decision made to prescribe ADT (Degarelix or LHRH agonist) prior to enrolment

Exclusion Criteria:

* Patient had previous or is currently under hormonal management of Prostate Cancer, except for a curative intention, where the duration of the neoadjuvant/adjuvant therapy did not exceed 6 months and treatment should have been terminated at least 6 months prior to baseline.
* Participation in a clinical trial at baseline and during the follow-up period

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced prostate cancer where a treatment decision on therapy has already been made according to medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Level of urologist's knowledge of patients' medical history at the point of decision making and during Androgen Deprivation Therapy (ADT) | Up to 4 years
  Measured by questionnaires by quantifying the frequency of urologists' entries
Level of urologist's knowledge of patients' comorbidities at the point of decision making and during ADT | Up to 4 years
  Measured by questionnaires by quantifying the frequency of urologists' entries
Level of urologist's knowledge of patients' concomitant medications at the point of decision making and during ADT | Up to 4 years
  Measured by questionnaires by quantifying the frequency of urologists' entries
Level of urologist's knowledge of patients' risk factors at the point of decision making and during ADT | Up to 4 years
  Measured by questionnaires by quantifying the frequency of urologists' entries

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational site (there may be other sites in this country), Rottweil, Germany

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976